CLINICAL TRIAL: NCT06446960
Title: The Role of Peripheral Afferents in Modulating Post-stroke Central Pain
Acronym: APEDOC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C23-05; 2023-504676-17-00 (Other: N° EU CT)
Record Dates: First submitted 2024-01-30; First posted 2024-06-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Ischemic Stroke; Central Neuropathic Pain
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Lidocaine; Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to receive one of 3 study treatments (lidocaine 20 mg/ml, levobupivacaine 1.25 mg/ml, or saline).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It is a randomised, double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lidocaine 20 mg/ml (Experimental): Name (INN and/or speciality) : Lidocaine 20 mg/ml Pharmaceutical form: Injectable Route of administration: Peri-Nervous Dosage for administration: 20ml Duration of treatment: 2 bolus administrations at 14 day intervals
  Interventions: Drug: Lidocaine 20mg/ml
- levobupivacaine 1.25 mg/ml (Experimental): Name (INN and/or speciality) : Levobupivacaine (Chirocaine), 1.25 mg/ml Pharmaceutical form: Injectable Route of administration: Peri-Nervous Dosage for administration: 20ml Duration of treatment: 2 bolus administrations at 14 day intervals
  Interventions: Drug: Levobupivacaine Hydrochloride 1.25 MG/ML
- Sodium chloride (NaCl) 0.9 (Placebo Comparator): Name (INN and/or speciality) : Sodium chloride (NaCl) 0.9 Pharmaceutical form: Injectable Route of administration: Peri-Nervous Dosage for administration: 20ml Duration of treatment: 2 bolus administrations at 14 day intervals
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Lidocaine 20mg/ml — 2 bolus administrations at 14 day intervals Route of administration: Peri-Nervous Dosage for administration: 20ml
  Arms: lidocaine 20 mg/ml
Drug: Levobupivacaine Hydrochloride 1.25 MG/ML — 2 bolus administrations at 14 day intervals Route of administration: Peri-Nervous Dosage for administration: 20ml
  Arms: levobupivacaine 1.25 mg/ml
Drug: Sodium Chloride 0.9% Inj — 2 bolus administrations at 14 day intervals Route of administration: Peri-Nervous Dosage for administration: 20ml
  Arms: Sodium chloride (NaCl) 0.9

SUMMARY:
Central post-stroke pain (CPP) is extremely difficult to relieve and responds very poorly to analgesics targeting neuropathic pain, probably because the mechanisms underlying this pain remain poorly understood.

Stroke pain is traditionally considered to be of central origin and related to changes in the spinal cord and/or brain nociceptive systems. However, a recent study in a small cohort of patients has suggested that the peripheral nervous system (PNS) may have a role in the initiation and persistence of APD.

The main objective of this prospective randomised controlled bicentric study (Raymond Poincaré and Ambroise Paré) in double blind and parallel groups against placebo (3 arms) will be to evaluate the efficacy of two peripheral nerve blocks performed 14 days apart on spontaneous neuropathic pain after stroke. The active treatments used for the blocks will be either lidocaine 20 mg/ml or levobupivacaine 1.25 mg/ml or placebo (saline)

DETAILED DESCRIPTION:
The primary endpoint will be the change in neuropathic pain intensity (assessed on an 11-point pain intensity scale), expressed as a difference in pain intensity between the value obtained before each block and that obtained 45 minutes after, corresponding to the maximum expected effect. Secondary endpoints will include exertional pain, pain quality, % relief, clinical global impression, pain assessment on a patient diary for a fortnight after each block and adverse events.

Patients will be randomised to receive one of 3 study treatments (lidocaine 2%, levobupivacaine 1.25 mg/ml or placebo). The treatment protocol will involve 2 perineural blocks performed 14 days apart. Assessment will continue for up to 2 weeks after each block, i.e. up to one month after the start of treatment. An evaluation of pain will be carried out before the block and after each block, at 45 minutes and at 5 hours, and then daily by the patient on a self-evaluation booklet for the 14 days following each block.

Randomisation will be centralised on a server from a list drawn up in advance by computer rogramme, balanced by blocks of variable size. Allocation between the 3 arms will be done according to a balanced 1:1:1 distribution. Treatments will be numbered from 1 to n, and allocated to patients in the chronological order of their inclusion in the trial.

Patients will be randomised on the day of treatment using a centralised computerised randomisation procedure to receive one of the 3 study treatments (lidocaine 20 mg/ml levobupivacaine 1.25 mg/ml or saline). No matching by age or duration of pain is planned, as randomisation usually results in groups matched at baseline on these criteria. The treatment will be administered over two visits performed 14 days apart by a qualified anaesthetist using the peri-nervous route according to current ecommendations (see above). Only one randomisation will be performed at baseline, so that a patient on active treatment cannot receive placebo at a later date and vice versa (see figure 1).

The investigators plan to randomise 10 patients per group and a total of 30 patients to achieve 90% power with a two sided α risk=0.05,. Given the estimated premature discontinuation rate, the investigators consider it necessary to include 12 patients per group for a total of 36 patients.

This study opens the way to new therapeutic avenues for these patients who often fail all treatments

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and over with no maximum age (blocks are generally very well tolerated in the very elderly)
2. Pain in the upper or lower limb distal enough to be completely covered by a peripheral nerve block
3. Chronic pain for at least 6 months
4. Ischaemic or haemorrhagic stroke for at least 6 months documented clinically and by appropriate imaging (MRI)
5. Post-stroke central neuropathic pain defined as pain occurring in the aftermath of stroke meeting the criteria for probable or defined neuropathic pain according to the NeuPSIG algorithm and with a DN4 screening questionnaire score of at least 4 out of 10.
6. Spontaneous pain intensity greater than or equal to 4 out of 10 on an 11-point numerical scale (EN) at inclusion and randomisation (i.e. just before each block)
7. Patients affiliated to a social security scheme or beneficiaries of such a scheme
8. Stable oral analgesic pharmacological treatment for at least 2 weeks prior to inclusion
9. Acceptance and signing of the informed consent

Exclusion Criteria:

1. Inability or unwillingness to sign an informed consent
2. Person subject to a legal protection measure (safeguard of justice, curatorship, guardianship)
3. Patients with ongoing psychiatric pathology (major depression, psychosis) or cognitive disorders that prevent a good understanding of the protocol and questionnaires
4. Pain that is too widespread in one hemicycle or limb and cannot be adequately covered by blocks
5. Ongoing drug or substance abuse
6. Language (aphasia) or comprehension disorders, illiteracy
7. Moderate to severe renal or hepatic impairment
8. Contraindication to local anaesthetics for use in perineural blocks (infection or acute inflammation in the injection area, known allergy).
9. Pregnancy or breastfeeding
10. Known hypersensitivity to lidocaine, levobupivacaine, amide-linked local anaesthetics or to any of the excipients contained in the specialities used in the study.
11. Patients with recurrent porphyria or severe hypotension contraindicating treatment with lidocaine and/or levobupivacaine
12. Current treatment with antiarrhythmic drugs causing torsades de pointes (amiodarone, disopyramide, quinidinics, sotalol...) or with antiarrhythmic drugs with local anaesthetic activity (mexiletine or class III antiarrhythmic drugs) and cannot be discontinued.
13. Too little pain at the time of the blocks (< 4 out of 10)
14. Need to modify analgesic pharmacological treatment at the beginning or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of two peripheral nerve blocks performed 14 days apart on spontaneous neuropathic pain after stroke. The active treatments used for the blocks will be either lidocaine 20mg/ml or levobupivacaine 1.25mg/ml or placebo (saline) | 24 months
  The evolution in neuropathic pain intensity assessed on an 11-point pain intensity scale (0 = no pain: 10: maximum imaginable pain), expressed as a difference in pain intensity between the value obtained before each block and that obtained 45 minutes after, corresponding to the maximum expected effect. The values obtained before and after each block will first be analysed individually and then combined for the two successive blocks for each patient and the comparison will be between the three treatment arms, lidocaine 20mg/ml, levobupivacaine 1.25mg/ml or placebo
  Rationale for the choice of the main criterion :
  Pain intensity will be assessed on a numerical scale that corresponds to the usual validated measurement criterion and the choice of 45 minutes corresponds to the maximum effect of local anaesthetics

SECONDARY OUTCOMES:
- To evaluate the time course and duration of the effectiveness of the nerve blocks on spontaneous pain on a pain intensity scale completed daily by the patient on a self-evaluation booklet up to 14 days after each block. | 24 months
  - Comparison of the duration (in days) of efficacy of lidocaine 20 mg/ml levobupivacaine 1.25 mg/ml and placebo blocks on spontaneous and exertional pain assessed by an 11-point pain intensity scale (0 to 10) completed daily by the patient on a self-report diary, up to 14 days after each block.
- Evaluate the effectiveness of blocks on exercise pain | 24 months
  - Comparison of the efficacy of levobupicacaine 1.25 mg/ml, lidocaine 20 mg/ml and placebo on spontaneous and exertional pain assessed by an 11-point pain intensity scale (0 to 10) at 45 minutes and then at 5 hours after the block and then daily on a self-evaluation booklet, up to 14 days after each block
- Directly compare the efficacy of active blocks, i.e. lidocaine and levobupivacaine, on spontaneous and provoked pain (allodynia) | 24 months
  * Comparison of the efficacy of lidocaine, levobupivacaine and placebo blocks on the intensity of rubbing pain if present (dynamic mechanical allodynia) assessed before treatment with a brush and then at 45 minutes and at 5 hours after each block.
  * Comparison of the efficacy of lidocaine, levobupivacaine and placebo blocks on spontaneous and provoked pain area (mechanical allodynia if present) assessed by a tracing (and then plotted on a graph allowing measurement of area in cm2) before treatment and then at 45 minutes and at 5 hours after each block using a method used in our previous studies
- Evaluate the effectiveness of each block on provoked pain (mechanical allodynia), mechanical, hot and cold pain thresholds and pain area | 24 months
  - Comparison of the efficacy of lidocaine, levobupivacaine and placebo blocks on mechanical pain and detection thresholds assessed by Semmes Weinstein monofilaments (calibrated from 0.057 g to 300 g) as well as on thermal pain and detection thresholds assessed by a thermotest before the treatment and at 45 minutes and at 5 hours after each block
- Evaluate the effectiveness of each block on the dimensions of neuropathic pain assessed by the NPSI questionnaire | 24 months
  - Comparison of the efficacy of lidocaine, levobupivacaine and placebo blocks on dimensions of neuropathic pain assessed by the NPSI questionnaire before treatment and at 45 minutes, and at 5 hours and 2 weeks after each block
- To evaluate the effectiveness of the blocks on the overall clinical impression, the percentage of relief as well as the satisfaction with the treatment | 24 months
  Evaluation of adverse effects of lidocaine, levobupivacaine and placebo blocks after the blocks and up to 14 days after each block.
  * Efficacy of lidocaine, levobupivacaine and placebo blocks on patient (PGIC) and examiner (CGIC) clinical global impression at 45 minutes, and at 5 hours and 2 weeks after each block.
  * Proportion of responders to lidocaine, levobupivicaine and placebo treatments assessed at 45 minutes, ad at 5 hours and 2 weeks after each block.
- Assessing the adverse effects of each treatment | 24 months
  - Evaluation of adverse effects of lidocaine, levobupivacaine and placebo blocks after the blocks and up to 14 days after each block
- Assessing the maintenance of blinding by a blinding questionnaire at the end of the study | 24 months
  - Blinding assessment by a blinding questionnaire at the end of the study for each patient

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Ambroise Paré, Boulogne-Billancourt
  - Hôpital Raymond Poincaré, Garches

IPD SHARING:
Plan to Share IPD: No